CLINICAL TRIAL: NCT06053255
Title: Safety and Efficacy of the Neurolyser XR for the Treatment of Low Back Pain Related to Sacroiliitis
Brief Title: Use of the Neurolyser XR for the Treatment of Low Back Pain Related to Sacroiliitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: FUSMobile Inc. (Industry)
Collaborators: Focused Ultrasound Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIJ-002
Record Dates: First submitted 2023-09-06; First posted 2023-09-25 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Sacroiliitis
Keywords: neurolysis; high-intensity focused ultrasound; nerve ablation; neurotomy; sacral joint pain
MeSH Terms: conditions — Sacroiliitis

STUDY DESIGN:
Intervention Model Description: 10 participant feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- HIFU for Sacroiliitis (Experimental): High-intensity focused ultrasound delivered to the lateral sacral branch nerve for neurolysis.
  Interventions: Device: High-intensity focused ultrasound for Sacroiliitis using the Neurolyser XR

INTERVENTIONS:
Device: High-intensity focused ultrasound for Sacroiliitis using the Neurolyser XR — HIFU is delivered via a non-invasive ultrasonic transducer, through a gel pad for acoustic coupling, into the patients body in a precise manner focused on the lateral sacral branch nerves.

SUMMARY:
The Neurolyser XR is a device used to deliver high-intensity focused ultrasound for the ablation of the lateral sacral branch nerve in patients with Sacroiliitis.

DETAILED DESCRIPTION:
The sacroiliac joint connects the sacrum (a triangle shaped bone) with the iliac bone on both sides of the lower spine. These joints transmit all the forces from the upper body to the pelvis and their respective legs. Repeated trauma and aging affect this joint resulting in inflammation and arthritic changes. These changes result in misalignment of the joint or limitation to normal motion which can create pain typically very low in the back or in the buttocks,

High-Intensity Focused Ultrasound (HIFU) technology uses sound waves. These sound waves are concentrated into a specific spot in order to raise the local tissue temperature causing a burn, this burn is expected to intentionally damage the nerve causing pain.

The HIFU device used in this study is called, the Neurolyser XR. It focuses sound wave energy directly on the nerve of the painful sacroiliac joint, causing an increase in temperature, which is expected to directly damage the nerve fibers which carry pain signals to the brain.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 and older
2. BPI < 40
3. Patients who are able and willing to give consent and able to attend all study visits.
4. Patients who are able to communicate with the treating physician.
5. Patients must have chronic lower back pain (LBP) attributed to degenerative sacroiliitis diagnosed by a pain physician using the following guidelines:
6. At least 1 positive sacroiliac joint provocation test (Gaeslen's test, FABER (Patrick's test), and pelvic rock)
7. Back pain predominantly below L5
8. 50% relief following either sacroiliac joint (SI) joint injection and/or lateral branch blocks corresponding to the expected duration of the medication utilized. (i.e SI joint injection-expected pain relief duration of steroid, lateral branch blocks-expected pain relief duration of local anesthetic utilized).
9. All other possible sources of low back pain have been ruled out as the primary pain generator, including but not limited to: the intervertebral discs, bone fracture, the zygapophyseal joints, the hip joint, symptomatic spondylolisthesis, tumor, and other regional soft tissue structures (this is done by physical exam, medical history, and MRI/CT/X-ray as required)
10. Patients with NRS (0-10 scale) LBP average score ≥ 4
11. Patients with chronic LBP for at least 12 months.
12. Patients with Oswestry Disability Questionnaire (ODQ) for LBP score > 40%

Exclusion Criteria:

1. Patients on dialysis
2. Patients with evidence of lumbosacral radiculopathy on MRI, CT or physical exam findings, including radicular leg pain (symptomatic moderate or severe foraminal or central canal stenosis).
3. Spinal pathology that may impede recovery such as spina bifida occulta, grade II or higher.
4. Spondylolisthesis at L5/S1, or scoliosis
5. Patients with radiofrequency ablation (RF/RFA) treatment for sacroiliitis LBP
6. Patients with bilateral sacroiliitis LBP
7. Patients with previous low back surgery
8. Patients who are pregnant
9. Patients with existing malignancy
10. Patients with allergies to relevant anesthetics
11. Patients with motor deficit or any other indication for surgical intervention
12. Patients with contraindications for MRI
13. Patients with an acute medical condition (e.g., pneumonia, sepsis, systemic infection, uncontrolled immunosuppression-AIDS, cancer, DM) that is expected to hinder them from completing this study.
14. Patients with unstable cardiac status including:
15. Unstable angina pectoris on medication
16. Patients with documented myocardial infarction less than 40 days prior to protocol enrolment
17. Patients with Severe Congestive Heart Failure, New York Heart Association (NYHA) class 4.
18. Patients on anti-arrhythmic drugs or with uncontrolled and/or untreated arrhythmia status
19. Patients with severe cerebrovascular disease (CVA within last 6 months)
20. Patients with severe hypertension (diastolic BP > 100 on medication)
21. Patient Body Mass Index > 45 or <20
22. Patients with known intolerance or allergies to the MRI contrast agent (e.g. Gadolinium or Magnevist) including advanced kidney disease
23. Patients with an active infection or severe hematological, neurological, or other uncontrolled disease.
24. The patient is unable to communicate with the investigator and staff.
25. Patients who are not able or willing to tolerate the required prolonged stationary position during treatment (approximately 2 hours)
26. Patient with acute pelvic inflammatory conditions
27. Ongoing/ unresolved Worker's compensation, injury litigation, military medical board, or disability remuneration claims
28. Morphine Milligram Equivalents (MME) > 60 per 24 hrs.
29. Patients with platelets < 100.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
The number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v6.0. | Procedure through 6 month follow-up visit
  Per the CTCAE assessment, each organ or possible adverse event would be categorized on a scale of 1 to 5 where:
  Grade 1 is Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 is Moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL).
  Grade 3 is Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL.
  Grade 4 is Life-threatening consequences; urgent intervention indicated. Grade 5 is Death related to AE.

SECONDARY OUTCOMES:
The participants change in level of pain as assessed by the Numerical Rating Scale (NRS) and any change in analgesic/opiate usage. | Procedure through 6 month follow-up visit
  The pain scale is 0 to 10 where 0 is no pain at all and 10 is the worst pain imaginable
Change in quality of life will be assessed by Oswestry Disability Index (ODI) | Procedure through 6 month follow-up visit
  ODI scale includes 10 questions, each can score 0 to 5 for a total score of 0 to 50.
  scores are interpreted as follows: 0-4: No disability 5-14: Mild disability 15-24: Moderate disability 25-34: Severe disability 35-50: Completely disabled
Change in quality of life will be assessed also by Brief Pain Inventory (BPI-QOL) | Procedure through 6 month follow-up visit
  BPI includes 7 questions on the level the patient pain interferes with their daily activities.
  Each question can score 0 to 10 for a total score of 0 to 70.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Kohan, MD, Principal Investigator — University of Virginia Pain Medicine Clinic
Locations (1):
- University of Virginia, Department of Anesthesiology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perez J, Gofeld M, Leblang S, Hananel A, Aginsky R, Chen J, Aubry JF, Shir Y. Fluoroscopy-Guided High-Intensity Focused Ultrasound Neurotomy of the Lumbar Zygapophyseal Joints: A Clinical Pilot Study. Pain Med. 2022 Jan 3;23(1):67-75. doi: 10.1093/pm/pnab275. PMID 34534337